CLINICAL TRIAL: NCT07244237
Title: Validity of an AI-Supported Whole-Body Electrical Stimulation Device for Spinal Pain Assessment: A Comparison With Self-Reported Pain Scores
Brief Title: Assessing Spinal Pain With an Artificial Intelligence-assisted Whole Body Electrical Stimulation Device
Status: Recruiting | Type: Observational
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Kübra Okuyucu, Associate Professor, Amasya University
Other Study IDs: 14082025
Record Dates: First submitted 2025-08-15; First posted 2025-11-24 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chronic Back Pain
Keywords: StimaWELL 120MTRS system; Chronic Back Pain; Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic back pain

SUMMARY:
The goal of this observational study is to investigate the correlation between self-reported pain and the measurements obtained using an artificial intelligence-assisted whole-body electrical stimulation device (StimaWELL 120MTRS system) in individuals with chronic back pain. The main question it aims to answer is: Is there any correlation between the pain intensity assessed with StimaWELL 120MTRS system, dolorimeter and self-report in adults with chronic back pain? The patients who have back pain for the duration longer than 3 months and have been eximaned by a medical doctor will be assessed with StimaWELL 120MTRS system, dolorimeter, and will be asked to rate their pain intensity in Numerical Pain Rating Scale.

DETAILED DESCRIPTION:
The goal of this observational study is to investigate the correlation between self-reported pain and the measurements obtained using an artificial intelligence-assisted whole-body electrical stimulation device (StimaWELL 120MTRS system) in individuals with chronic back pain. This study is designed as an exploratory, cross-sectional study. After obtaining written and verbal informed consent, 200 patients with back pain will be asked about their age, sex, height, weight, and duration of back pain. Pain location and intensity will be assessed by one of the investigators using a body diagram and the Numerical Pain Rating Scale (NPRS). In addition, the patients will be evaluated by another investigator using the StimaWELL 120MTRS device, and using the dolorimeter for the pressure pain threshold (PPT). PPT will be assessed at four bilateral points: the upper trapezius, the lower trapezius, 5 cm lateral to the spinous process of the L3 vertebra, and 2 cm cranial to the posterior superior iliac spine. To achieve 80% power at a 5% significance level, assuming a medium effect size, estimated minimum sample size is calculated as 158 participants. Accordingly, the target sample size is set at 200 participants. Pearson's or Spearman's correlation coefficient will be used to determine the relationship between pain values measured by the artificial intelligence-assisted device and patient-reported pain scores (0-10) or pressure pain threshold. To assess the relationships among the three continuous variables obtained in this study-patient-reported pain scores (0-10), device-measured pain values, and pressure pain threshold-repeated-measures ANOVA or the Friedman test will be used to compare their means.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing back pain for more than three months
* Experiencing recurrent back pain over the last week
* Not having used analgesic or muscle relaxant medications in the last week
* Aged between 18 and 60 years
* Diagnosed with chronic low back pain by a medical doctor
* Literate and able to cooperate with study procedures
* Willing to participate in the study

Exclusion Criteria:

* Having neurological, inflammatory, radiculopathy, vertebral fracture, or similar conditions
* Experiencing acute-onset pain
* Being pregnant or at risk of pregnancy
* Having a psychiatric diagnosis and currently taking medication
* Having a skin disease or lesion in the area where electrodes will be applied
* Currently undergoing physical therapy
* Having vestibular, auditory, or cognitive impairments
* Possessing an electronic implant
* Having a cardiac arrhythmia
* Having a coronary or carotid stent
* Being diagnosed with epilepsy
* Having severe osteoporosis of the spine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be recruited from the eligible and volunteer patients who will visit the healthy living center in study duration.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Pain intensity measured by the StimaWELL 120MTRS system | baseline, one time
  The StimaWELL® EMS device is a high-tech modulated low-frequency, 12-channel, mid-frequency stimulation device. The output of the calibration process will be recorded as data to use in the analysis.
Pressure pain threshold | baseline, pre-procedure
  PPT will be assessed using a dolorimeter at four bilateral points (upper trapezius, lower trapezius, 5 cm lateral to L3 spinous process, and 2 cm cranial to the posterior superior iliac spine).
Patient-reported pain | baseline, pre-procedure
  Participants will be asked to indicate the location of their back pain experienced over the last week on a body diagram, which shows the regions where the electrodes will be placed in a faint outline. For each marked region, participants will be asked to rate their pain intensity using the Numerical Pain Rating Scale. The scale ranges from 0 to 10, where 0 indicates "no pain" and 10 indicates "worst imaginable pain." Higher scores represent greater pain intensity.

CONTACTS AND LOCATIONS:
Locations (1):
- AMASYAŞAM Sağlıklı Yaşam Merkezi, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
IPD will probably be shared on a reasonable request. But it is not decided yet.